CLINICAL TRIAL: NCT04776213
Title: A 2-year Follow-up Study to Assess Cognition and Health-related Quality of Life in Participants With Highly-active Relapsing Multiple Sclerosis, Having Participated in the CLARIFY MS Trial (CLARIFY MS Extension)
Brief Title: Cognition and HRQoL in Adults With Highly-active RMS in Year 3 and 4 After Initial Mavenclad® Dose (CLARIFY MS Extension)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MS700568_0158; 2020-003874-30 (EudraCT Number)
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Health related quality of life; Mavenclad®; Relapsing Multiple Sclerosis; Cladribine; Cognitive impairment cognition; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mavenclad® (Experimental)
  Interventions: Drug: Mavenclad®

INTERVENTIONS:
Drug: Mavenclad® — This low interventional extension study involves the follow up of participants in the parent study. The participants were followed up for an additional 2 year period (until 4 years after initial administration of Mavenclad® tablets), during which the participants were not treated with Mavenclad®, as per European Medicines Agency (EMA) label of Mavenclad®.

SUMMARY:
The purpose of the study was the evaluation of the effect of a treatment for highly-active relapsing multiple sclerosis (RMS). This was the extension study to CLARIFY MS (NCT03369665), to assess cognitive impairment and health related quality of life (HRQoL) in participants with highly active RMS, at 4 years after initial dose of Mavenclad® tablets.

ELIGIBILITY:
Inclusion Criteria:

* Have at least CLARIFY MS Baseline data on Symbol Digit Modalities Test (SDMT)
* Received at least a single dose of cladribine tablets in the CLARIFY MS study
* Completed the Final Study Visit (M24) of the CLARIFY MS study
* Capable of giving signed informed consent, as indicated in protocol, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and this protocol

Exclusion Criteria:

* Participant is considered by the Investigator and Sponsor, for any reason, to be an unsuitable candidate for the study
* Participation in other studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (60):
- Eva Maida, Vienna, Austria
- Czechia (8):
  - FN u sv. Anny Brno, Brno
  - FN Hradec Králové, Hradec Králové
  - Nemocnice Jihlava, p.o., Jihlava
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava
  - Faculty Hospital Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Nemocnice Teplice, Teplice
- Denmark (2):
  - Glostrup Sygehus, Glostrup Municipality
  - Odense Univeristy Hospital, Odense
- France (10):
  - Centre hospitalier de la Côte Basque - Saint Léon, Bayonne
  - Pellegrin, Bordeaux
  - CHU de la Côte de Nacre, Caen
  - Centre Hospitalier de Gonesse, Gonesse
  - CHRU de Lille Hôpital Roger Salengro, Lille
  - CHU Hôpital Nord Laennec, Nantes
  - Hôpital de la Pitié-Salpétrière, Paris Cédex 13
  - CHU de Poissy, Poissy
  - Centre Universitaire de Rouen, Rouen
  - CHU Tours - Hôpital Bretonneau, Tours
- Hungary (6):
  - Jahn Ferenc Dél-Pesti Kórház és Rendelőintézet, Budapest
  - Semmelweis University II, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum, Debrecen
  - Valeomed Kft, Esztergom
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókór, Nyíregyháza
- Italy (13):
  - A.O.U. Ospedali Riuniti Umberto, Ancona
  - University of Cagliari, Cagliari
  - PO G.Rodolico, AOU Policlinico-Vittorio Emanuele Catania, Catania
  - Ospedale San Raffaele Giglio, Cefalù
  - Instituto Nazionale Neurologico "Carlo Besta", Milan
  - Ospedale San Raffaele, IRCCS, Milan
  - A.O. Universitaria Federico II, Napoli
  - Policlinico Università della Campania L. Vanvitelli, Napoli
  - A.O. Ospedali Riuniti Villa Sofia-Cervello U.O. Endocrinolog, Palermo
  - Azienda Ospedaliera S. Camillo Forlanini, Roma
  - Neurological Center of Latium, Roma
  - Ospedale Sant'Andrea Neurologia - Università La Sapienza, Roma
  - Policlinico Tor Vergata, Roma
- Zuyderland, Sittard-Geleen, Netherlands
- Poland (7):
  - COPERNICUS Podmiot Leczn. Sp z o.o., Gdansk
  - M.A.-Lek A.M. Maciejowscy S.C. Centrum Terapii SM, Katowice
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Uniwersytecki Szpital Kliniczny nr 1 i.m. Norberta Barlickie, Lodz
  - Indywidualna Praktyka Lekarska Prof. Konrad Rejdak, Lublin
  - Centrum Medyczne Medyk, Rzeszów
  - Instytut Psychiatrii i Neurologii - Dept of Neurology II, Warsaw
- Slovakia (4):
  - Neuropoint s.r.o, Bratislava
  - Univerzitna nemocnica Martin, Martin
  - Fakultna nemocnica Nitra, Nitra
  - Fakultna nemocnica Trnava, Trnava
- Spain (8):
  - Hospital Universitario de Getafe, Getafe
  - C.A.U. de León - H. de León, León
  - Hospital Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan Despí
  - Hospital Universitario Nuestra Senora de la Candelaria, Santa Cruz de Tenerife
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0158
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 280 participants were enrolled in the study from different study sites.
Groups:
- Mavenclad®: This low interventional extension study involves the follow up of participants in the parent study (NCT03369665). The participants were followed up for an additional 2 year period (until 4 years after initial administration of Mavenclad® tablets), during which the participants are not treated with Mavenclad®, as per European Medicines Agency (EMA) label of Mavenclad®.
Period: Overall Study
Arm/Group | Mavenclad®
Started | 280
Completed | 269
Not Completed | 11
Not completed — Other | 1
Not completed — Withdrawal by Subject | 7
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all eligible participants, for whom any Visit data had been collected after end date of CLARIFY MS Year 2 Visit (Month 24 Visit).
Arm/Group | Mavenclad®
Number analyzed (Participants) | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201
  Male | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 202
  Unknown or Not Reported | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 248
  More than one race | 0
  Unknown or Not Reported | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With No or Minimal Decline in Cognitive Function, Defined As an Improved or Stable Symbol Digit Modalities Test (SDMT) Score or a Decline of 4 Points or Less in the SDMT Score, From Baseline of Parent Study to Month 48
Description: The SDMT is a test of information processing speed. It consists of 9 abstract symbols. Each symbol is paired with a single digit. The participant is provided with a "key", showing each symbol digit pair. In addition, the participants are shown several rows of the 9 symbols, which are arranged pseudo-randomly, without the digit. Participants are asked to voice the digit associated with each symbol as rapidly as possible for 90 seconds. The SDMT score ranges from 0 to 110 where higher scores indicated improvement and lower scores indicated worsening.
Time Frame: Baseline (Baseline of parent study [NCT03369665]) and Month 48 after initial dose of Mavenclad® in parent study (NCT03369665)
Population: Full analysis set (FAS) included all eligible participants, for whom any Visit data had been collected after end date of CLARIFY MS (NCT03369665) Year 2 Visit (Month 24 Visit).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mavenclad®
Number analyzed (Participants) | 280
percentage of participants | 68.6 [62.9 to 73.7]

2. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQoL) as Measured by Multiple Sclerosis Quality of Life 54 Questionnaire (MSQoL-54) Physical and Mental Health Composite Summary Scores at 4 Years
Description: The MSQOL-54 was a multidimensional health-related QOL measure that combines both generic and MS-specific items into a single instrument. This 54-item instrument generates 12 sub-scales along with two summary scores, and two additional single-item measures. Sub-scales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The two summary scores physical health and mental health are derived from a weighted combination of scale scores. Each composite summary score has a range from 0-100 where higher scores indicate better QOL. A positive change from baseline indicates improvement.
Time Frame: Baseline (baseline of parent study [NCT03369665]), 4 years after initial dose of Mavenclad® in parent study (NCT03369665)
Population: Full analysis set (FAS) included all eligible participants, for whom any Visit data had been collected after end date of CLARIFY MS (NCT03369665) Year 2 Visit (Month 24 Visit). Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mavenclad®
Number analyzed (Participants) | 265
score on a scale
  Physical health composite score | 3.69 [1.71 to 5.67]
  Mental health composite score | 5.13 [2.73 to 7.53]

3. Secondary Outcome: Change From Month 24 in Health Related Quality of Life (HRQoL) as Measured by Multiple Sclerosis Quality of Life 54 Questionnaire (MSQoL-54) Physical and Mental Health Composite Summary Scores at 4 Years
Description: as for outcome 2
Time Frame: Month 24 after initial dose of Mavenclad® in parent study (NCT03369665), 4 years after initial dose of Mavenclad® in parent study (NCT03369665)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mavenclad®
Number analyzed (Participants) | 232
score on a scale
  Physical health composite score | -2.02 [-3.81 to -0.22]
  Mental health composite score | -0.36 [-2.65 to 1.92]

ADVERSE EVENTS:
Time Frame: Up to 4 years after initial dose of Mavenclad® in parent study (NCT03369665).
Arm/Group | Mavenclad®
All-Cause Mortality (participants affected / at risk) | 0/280
Serious Adverse Events (participants affected / at risk) | 15/280
Other Adverse Events (participants affected / at risk) | 110/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mavenclad® (N=280)
Diverticulum intestinal (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Bartholin's abscess (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Loss of consciousness (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Stress urinary incontinence (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mavenclad® (N=280)
COVID-19 (Infections and infestations) | 84
Headache (Nervous system disorders) | 21
Nasopharyngitis (Infections and infestations) | 16
Urinary tract infection (Infections and infestations) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT04776213/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT04776213/SAP_001.pdf